CLINICAL TRIAL: NCT01085721
Title: Comparison Between Dexchlorpheniramine and Dexchlorpheniramine/Pseudoephedrine/Guaifenesin in the Relief of Allergic Symptoms in Rhinitic Patients With Viral Upper Respiratory Tract Infections and Productive Cough
Brief Title: Comparison Between Dexchlorpheniramine and Dexchlorpheniramine/Pseudoephedrine/Guaifenesin in Respiratory Infections
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mantecorp Industria Quimica e Farmaceutica Ltd. (Industry)
Responsible Party: Celso Pereira Sustovich, Medical Director, Mantecorp Indústria Química e Farmacêutica Ltda.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POE/P/09-1
Record Dates: First submitted 2010-03-09; First posted 2010-03-12 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Viral Infections of the Upper Respiratory Tract
Keywords: allergic rhinitis; viral infections of the upper respiratory tract; dexchlorpheniramine; pseudoephedrine; guaifenesin
MeSH Terms: conditions — Rhinitis, Allergic | interventions — dexchlorpheniramine; Pseudoephedrine; Guaifenesin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexchlorpheniramine pseudoephedrine guaifenesin (Experimental)
  Interventions: Drug: Dexchlorpheniramine, pseudoephedrine, guaifenesin
- Dexchlorpheniramine (Active Comparator)
  Interventions: Drug: Dexchlorpheniramine

INTERVENTIONS:
Drug: Dexchlorpheniramine, pseudoephedrine, guaifenesin — 5 mL (2 mg dexchlorpheniramine, 20 mg pseudoephedrine and 100 mg guaifenesin) qid for 5 days
  Arms: Dexchlorpheniramine pseudoephedrine guaifenesin
Drug: Dexchlorpheniramine — 5 mL (2 mg dexchlorpheniramine) qid for 5 days
  Arms: Dexchlorpheniramine

SUMMARY:
Patients with allergic rhinitis frequently present exacerbation of the atopic symptoms during viral infections of the upper respiratory tract. Also, allergic rhinitis makes the mucosa more reactive to infectious agents and potentiates mucus production.

The combination of dexchlorpheniramine, pseudoephedrine and guaifenesin elicits antihistaminic, decongestant and expectorant effects. The study hypothesizes is that this product is superior to dexchlorpheniramine alone in the relief of allergic symptoms and in promoting mucus elimination in atopic patients with viral infections of the upper respiratory tract.

ELIGIBILITY:
Inclusion Criteria:

* Patients with allergic rhinitis with symptoms of viral infection of the upper respiratory tract (rhinorrhea, nasal obstruction and productive cough)
* Compliance of the subject to the treatment protocol
* Agreement with the terms of the informed consent
* Patients who did not use forbidden medications

Exclusion Criteria:

* History of allergy to any component of the formulations
* Use of any investigational drug within the last 30 days
* Patients with bacterial infections of the upper respiratory tract
* Patients with high blood pressure (> 140 x 90 mmHg)
* Patients who are receiving inhaled beta-agonists or other antihistamine, decongestant or expectorant
* Patients with known pulmonary disease (asthma, COPD, neoplasias)
* Pregnancy
* HIV + patients
* Other conditions considered by the investigator as reasonable for non-eligibility

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)

PRIMARY OUTCOMES:
Symptoms frequency and intensity evaluated with a 5 point visual analogic scale (VAS) | 5 days

SECONDARY OUTCOMES:
Subjective evaluation of efficacy and tolerability graded as excellent, good, fair ou poor. | 5 days